CLINICAL TRIAL: NCT06135883
Title: Evaluating Folic Acid Awareness and Usage in High-Risk Pregnant Women for Neural Tube Defects
Brief Title: Assessing Folic Acid in High-Risk Pregnancy for Neural Tube Defects
Status: Completed | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Cagdas Nurettin Emeklioglu, MD, Karabuk University
Other Study IDs: KBU-EMEKLIOĞLU-001
Record Dates: First submitted 2023-11-08; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Neural Tube Defects; Folic Acid
Keywords: neural tube defects; folic acid; awareness; perinatology; pregnancy
MeSH Terms: conditions — Neural Tube Defects

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Singleton pregnant women over the age of 18 and under the age of 45 who have at least one of the risk factors for neural tube defects (family history, MTHFR gene mutation, birth history with aneuploidy, history of GDM or known DM).
- Control: Singleton pregnant women over 18 years of age and under 45 years of age who do not have any risk factors for neural tube defects

SUMMARY:
Aim of this study is to investigate and statistically reveal the prevalence and awareness of folic acid usage in pregnant women who have at least one of the risk factors for neural tube defects, to express the level of knowledge of the determined population on this subject and to present ideas to increase awareness in the society.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years
* Under 45 years of age
* Having at least one of the risk factors for neural tube defects (family history, MTHFR gene mutation, birth defect with aneuploidy, history of GDM or known DM) for Case Group.
* Singleton pregnant women

Exclusion Criteria:

* under 18 years old
* Above 45 years old
* Multiple pregnancies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Singleton pregnant women over the age of 18 and under the age of 45 who have at least one of the risk factors for neural tube defects (family history, MTHFR gene mutation, birth history with aneuploidy, history of GDM or known DM).
Sampling Method: Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
High awareness level for high-risk pregnant women | up to 12 weeks
  Pregnant women with at least one risk factor for neural tube defects have statistically higher folic acid use and awareness than control group pregnant women.
Low awareness level for society, regardless of the risk situation | up to 12 weeks
  Low folic acid knowledge and awareness in the sample groups, regardless of risk status

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Tascioglu City Hospital, Istanbul, Sisli, Turkey (Türkiye)